CLINICAL TRIAL: NCT03925714
Title: Investigating the Impact of p53 and SIRT1 in the Development of Type 2 DM Through the Treatment of Prediabetic Individuals by Either Nigetella Salivata or Metformin
Brief Title: Impact of P53 and SIRT1 in Type 2 Diabetes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: dm 2
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: DM
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- life style (Other): life style control only
  Interventions: Other: life style
- Metformin (Active Comparator): Metformin 500 mg twice daily
  Interventions: Drug: Metformin
- Nigetella salivata (Experimental): NS 450 mg twice daily
  Interventions: Drug: Nigetella salivata

INTERVENTIONS:
Other: life style — life sryle control only
  Other Names: life style management
  Arms: life style
Drug: Metformin — metformin twice daily
  Other Names: cidophage
  Arms: Metformin
Drug: Nigetella salivata — NS twice daily
  Other Names: NS
  Arms: Nigetella salivata

SUMMARY:
Investigating the impact of p53 and SIRT1 in the development of type 2 DM

DETAILED DESCRIPTION:
Investigating the impact of p53 and SIRT1 in the development of type 2 DM through the treatment of prediabetic individuals by either nigetella salivata or Metformin

ELIGIBILITY:
Inclusion Criteria:

* Prediabetic subjects.

Exclusion Criteria:

* Confirmed diabetes.
* Hepatic or renal impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improved insulin resistance | 6 months
  Number of patients showing improved insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Eman SA Sawan, Msc, Principal Investigator — Tanta University - Faculty of Pharmacy; Sahar Hegazy, Prof, Principal Investigator — Tanta University - Faculty of Pharmacy; Tarek Mostafa, ass. Prof., Study Director — Tanta University - Faculty of Pharmacy; Sherin El-Nidany, MD, Study Chair — Tanta University-Faculty of pharmacy
Locations (1):
- Sherief Abd-Elsalam, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mostafa TM, Hegazy SK, Elnaidany SS, Shehabeldin WA, Sawan ES. Nigella sativa as a promising intervention for metabolic and inflammatory disorders in obese prediabetic subjects: A comparative study of Nigella sativa versus both lifestyle modification and metformin. J Diabetes Complications. 2021 Jul;35(7):107947. doi: 10.1016/j.jdiacomp.2021.107947. Epub 2021 May 8. PMID 34006388